CLINICAL TRIAL: NCT02756143
Title: Exercise During Pregnancy and Perinatal Outcome. Randomized Controlled Trial
Brief Title: Exercise During Pregnancy and Perinatal Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Torrejon (Other)
Collaborators: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Maia Brik, MD PhD, University Hospital of Torrejon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PERINATEXER
Record Dates: First submitted 2016-04-21; First posted 2016-04-29 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Pregnancy; Healthy
Keywords: fetal heart; cesarean section; exercise; pregnancy
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Non- supervised physical exercise program during pregnancy
- Exercise Group (Experimental): Supervised physical exercise program during pregnancy
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Supervised physical conditioning program of three 55-60 minute sessions per week during whole pregnancy (from week 9 to 38). Each session consists of 25-30 minutes of cardiovascular exercise,10 minutes of specific exercises (strength and balance exercises), and 10 minutes of pelvic floor muscles training.
  Aerobic activity was prescribed at light to moderate intensity, aiming for 55-60% of heart rate reserve. All subjects wore a heart rate (HR) monitor (Polar FT7) during the training sessions to ensure that exercise intensity was light to moderate.
  Arms: Exercise Group

SUMMARY:
Effect of Physical Exercise Program on fetoplacental circulation and perinatal outcome.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of a supervised physical exercise program during pregnancy on fetoplacental circulation, fetal heart echocardiogram parameters and perinatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines
* Able to communicate in spanish
* Giving birth at Torrejon Universitary Hospital

Exclusion Criteria:

* Medical or obstetric complication excluding exercise ( ACOG guideline)
* Interested in the study after 18 weeks or pregnancy
* Not availability to attend to the physical exercise program

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Maternal weight gain during pregnancy | From the beginning of the pregnancy to 1 month postdelivery

SECONDARY OUTCOMES:
Cesarean Section Rate | Birth
Gestational Diabetes | Birth
Preeclampsia | birth
Fetal TAPSE | up to 36 weeks of pregnancy
  Tricuspid Annular Plane Systolic Excursion meassured by echocardiogram
Fetal Tei Index | up to 36 weeks of pregnancy
  Myocardial Performance Index meassured by echocardiogram
Ductus Arteriosus PI | up to 36 weeks
  Ductus Arteriosus Pulsatility Index meassured by echocardiogram
Aortic Isthmus PI | up to 36 weeks
  Aortic Isthmus Pulsatility Index meassured by echocardiogram
Fetal Heart Rate Variability | birth
  Fetal Heart Rate Variability meassured by cardiotocogram
Newborn weight | birth
  birth
Placental weight | birth

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Barakat, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- University Hospital de Torrejon, Torrejón de Ardoz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.youtube.com/watch?v=qlDs3pEp5Ro